CLINICAL TRIAL: NCT07386691
Title: Comparing Effect of Intradialytic Aerobic Exercise Versus Incentive Spirometer on Fatigue and Sleep Quality Among Hemodialysis Patients.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Haider Athab Mohammed, assist Lecturer, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BaghdadU Unique Protocol ID
Record Dates: First submitted 2026-01-21; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Fatigue; Sleep Disturbance; Hemodialysis Complication
Keywords: fatigue; sleep quality; Hemodialysis
MeSH Terms: conditions — Fatigue; Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial aims to compare the effects of intradialytic aerobic exercise versus incentive spirometer breathing exercises on fatigue and sleep quality among patients undergoing maintenance hemodialysis. Eligible participants will be randomly assigned to one of three parallel groups: intradialytic aerobic exercise, incentive spirometer intervention, or routine care (control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intradialytic aerobic exercise (Experimental): the best time for experimental is 30min after the initiation and during the first 2 h of dialysis . The researcher placed the bike on the bed, fixed the patient's feet to the pedals using adhesive straps, and knee range of motion was determined for each subject. Patients performed passive pedaling at low power for 20 min at a speed of 30rpm during the first 2h of every dialysis session. Participants were instructed on how to exercise and verbal encouragement was provided to them during exercise. Before, during, and after exercise, clinical assessment, blood pressure, heart rate and body temperature were obtained. If the participant had a blood pressure of 180/110 mmHg and higher, systolic pressure lower than 90mmHg, chest pain, shortness of breath, or high body temperature (> 37.8oC) before or during dialysis, the exercise would be discontinued. None of the patients suffered from such complications and all participated with out interruption.
  Interventions: Other: intradialytic aerobic exercise versus incentive spirometer
- Incentive Spirometer (Experimental): using incentive spirometer : - Loosen any tight clothing, especially around neck.
  * Each patient was instructed to sit upright with placing incentive spirometer at the same level of his mouth to promote optimal lung expansion while using the spirometer.
  * The patient was instructed to exhale letting all the breath out.
  * Ask the patient to close the lips around the mouthpiece of the spirometer.
  * Instruct the patient to inhale slowly, breathing in until unable to do any more, this would raise the balls to the top of the column.
  * Ask the patient to hold the breath as long as possible (at least five seconds) then exhale slowly.
  * Session was in the form of 30 times in sets, each set consist of 5-6 repetitions with rest 1 minute between sets.
  * Intensity of exercise was increased by increasing time of session, time of holding the breath and numbers of repetitions according to patient's status.
  * The training was 2 times/week for 4 weeks
  Interventions: Other: intradialytic aerobic exercise versus incentive spirometer
- control group (No Intervention): Routine care control group will not exposed to the intervention therapy and will take only routine care

INTERVENTIONS:
Other: intradialytic aerobic exercise versus incentive spirometer — The interventions were implemented during the first two hours of the hemodialysis session, starting 30 minutes after initiation. For intradialytic aerobic exercise, the cycle ergometer was placed on the bed, the patients' feet were secured to the pedals, and knee range of motion was assessed individually. pedaling was performed for 20 minutes at a speed of 30 rpm during each session, with instructions and verbal encouragement provided. Vital signs (blood pressure, heart rate, and body temperature) were monitored before, during, and after exercise.
  Regarding the use of the Incentive Spirometer, patients were seated upright and instructed to perform slow deep inhalation with breath holding for at least 5 seconds, followed by slow exhalation. Each session consisted of 30 repetitions divided into sets (5-6 repetitions per set) with a one-minute rest between sets. Exercise intensity was progressively increased according to the patient's condition. Training was conducted twice weekly
  Arms: Incentive Spirometer; intradialytic aerobic exercise

SUMMARY:
In order to accomplish the objectives of this investigation, a single-blind experimental comparative design was implemented to evaluate the impact of intradialytic aerobic exercise and Incentive Spirometer on sleep quality and fatigue. Three experimental groups (aerobic exercise and Incentive Spirometer) and one control group were subjected to pre- and post-tests. Is there a difference in the levels of fatigue and sleep quality between hemodialysis patients who receive aerobic exercise and incentive spirometer therapy and those who do not receive it? Researcher will compare the levels of fatigue and sleep quality between hemodialysis patients who receive interventional therapy and those who do not receive it to see if interventional therapy works to relieve the fatigue and improve sleep quality. Participants will take aerobic exercise therapy group applied on the leg muscles for 20 minutes per session, and incentive spirometer group on respiratory muscles

* Ask the patient to hold the breath as long as possible (at least five seconds) then exhale slowly.
* Session was in the form of 30 times in sets, each set consist of 5-6 repetitions with rest 1 minute between sets , 2 times per week for total one month, during the first hour of each hemodialysis. sessions.

DETAILED DESCRIPTION:
Irreversible loss of kidney function is known as chronic kidney failure, which can be fatal without dialysis or a kidney transplant . The incidence of chronic kidney disease (CKD) has been rising globally, leading to high rates of mortality, complications, and decreased quality of life. Currently, kidney problems affect more than 850 million people worldwide, and CKD is expected to rank fifth among the leading causes of premature death .

Dialysis is a common treatment for chronic kidney disease (CKD), which accounts for more than 89% of end-stage renal disease (ESRD) patients worldwide . Although dialysis prolongs life, it also leads to significant disabilities, including decreased physical capacity, reduced daily functioning, fatigue, reduced mobility, poor sleep quality, and deterioration in overall health . One of the most common and disabling complaints among dialysis patients is fatigue, which impairs their cognitive, physical, and psychological abilities. Patients frequently report reduced ability to perform daily tasks, persistent fatigue, increased daytime sleepiness, and impaired attention .

The prevalence of fatigue among dialysis patients ranged from 20% to 86% in a systematic review . Another common problem among dialysis patients is sleep disturbances, which significantly impact their quality of life. Poor sleep quality was reported by 68% of dialysis patients in a systematic review . Exercise is becoming increasingly important as a promising non-pharmacological treatment for improving heart and lung function in dialysis patients. Recent research suggests that physical activity enhances cardiovascular and physical function, as well as quality of life, in individuals undergoing maintenance dialysis. This leads to a positive cycle that includes improved mood, increased appetite, and increased food intake. Fatigue is defined as a persistent and severe state of tiredness that leads to mental or physical exhaustion, with a prevalence ranging from 60% to 97%. It is associated with a decreased quality of life and decreased survival rates . To recover, patients with post-dialysis fatigue must receive at least three hours of rest after each treatment session. Therefore, healthcare providers prioritize fatigue management as a treatment priority .Hemodialysis patients frequently experience sleep disturbances. The prevalence of sleep difficulties is estimated to range from 18% to 69%, with various forms, such as restless legs syndrome associated with obstructive sleep apnea. Sleep quality is the degree of satisfaction an individual feel with their sleep experience, which encompasses a variety of factors, including sleep rate, sleep duration, ability to stay asleep, and feeling refreshed upon awakening. Chronic fatigue, neurological changes, decreased self-care, and functional impairment are among the many problems that sleep deprivation can cause. Therefore, it is essential to prioritize sleep quality and address sleep deprivation in hemodialysis patients . A variety of pharmacological and non-pharmacological interventions can be beneficial for end-stage renal disease (ESKD) patients experiencing fatigue and sleep difficulties .

A symptom cluster forms when fatigue and sleep problems converge, meaning they frequently occur simultaneously and exacerbate each other. The quality of life and functional independence of dialysis patients is significantly impacted by managing this cluster, which is a therapeutic priority . Currently, limited pharmacological options are available to alleviate symptoms in this population. Side effects, interference with dialysis treatments, or inadequate relief are common consequences of medications. As a result, non-pharmacological interventions have become globally recognized as cost-effective, safe, and practical strategies. Deep breathing, mindfulness, relaxation techniques, and exercise are among the most widely researched approaches .

Clinical studies have demonstrated that aerobic exercise, particularly during dialysis, enhances dialysis efficiency, increases blood flow to muscles, removes toxins, and reduces inflammation . Aerobic exercise during dialysis has been shown to enhance cardiovascular function, reduce fatigue, and enhance overall health-related quality of life in clinical studies . Additionally, exercise can be performed during dialysis, as the patient does not need to spend a long period outside the dialysis center. Research has shown that deep breathing exercises are a beneficial complementary approach. Slow, purposeful breathing regulates the autonomic nervous system, increasing oxygenation, lowering blood pressure, and reducing sympathetic nervous system activity .

Visually feedback-based incentive spirometers aim to enhance respiratory muscle training and reverse and prevent lung disorders, leading to prolonged inspiratory duration and lung expansion dynamics. The combination of inspiratory pauses and sustained maximal inspiration increases trans pulmonary pressure, which negatively impacts lung inflation.

Nurses play a crucial role in assessing vital signs and managing pain, as they frequently and extensively interact with dialysis patients. Therefore, it is essential that they have the experience and skill to develop comprehensive nursing strategies specifically designed to address these concerns. Non-pharmacological techniques are frequently used in conjunction with pharmacological therapy to improve sleep quality and reduce fatigue during interventional procedures. Several studies have demonstrated the effectiveness of fatigue management during hemodialysis .

Researchers are currently investigating the effect of a variety of non-pharmacological methods on fatigue and sleep quality. However, no specific study has been conducted to compare and analyze the effects of incentive spirometry and aerobic exercise on sleep quality and fatigue in hemodialysis patients.

Research design In order to accomplish the objectives of this investigation, a single-blind experimental comparative design was implemented to evaluate the impact of intradialytic aerobic exercise and Incentive Spirometer on sleep quality and fatigue. Three experimental groups (aerobic exercise and Incentive Spirometer) and one control group were subjected to pre- and post-tests. Randomization guarantees analogous groups, mitigates selection bias, and facilitates causal inferences regarding the efficacy of an intervention.

Setting:

The research sample of hemodialysis patients will be served by the Al-Diwaniyah Government Hospital, which includes the Al-Hayat Dialysis Center, Fatima Al-Zahraa Dialysis Center, Afak General Hospital Dialysis Center, and Al-Shamiya General Hospital Dialysis Center in Diwaniyah, Iraq. The selection of these centers was based on the availability of patients and the fact that patients are treated according to a specific schedule during dialysis, which enables researchers to closely monitor their progress.

Sample and sampling:

To ensure a transparent and scientifically based randomization procedure, a probability (simple) sampling method was implemented to enroll patients in the study. sampling commences with the second random point of the scheduled patients who A study participant is represented by number one, while a non-study participant is represented by number two in a simple random sample. The participants were subsequently divided into three groups using simple random sampling. The patient was assigned to either the aerobic exercise, incentive spirometer, or control group by a sealed envelope containing three numbers: 1, 2, and 3. The patient was assigned to the aerobic exercise group, the incentive spirometer group, or the control group. Participants were unaware that aerobic exercise, incentive spirometer, and sleep quality were induced in hemodialysis patients, thereby ensuring the single-blind method was in place to prevent potential biases. In order to acquire data that is both accurate and representative, these two probability sampling methods were chosen.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-60 years
* Diagnosed with end-stage renal disease and receiving maintenance hemodialysis
* On hemodialysis for at least 3 months
* Experiencing fatigue and sleep disturbances
* Clinically stable during the study period
* Able to communicate and provide written informed consent

Exclusion Criteria:

* Unstable cardiovascular disease
* Severe musculoskeletal disorders limiting exercise
* Cognitive impairment
* Patients with diabetes mellitus for at least 10 years with diabetic neuropathy (DPN ≥ 6)
* Recent hospitalization within the last 4 weeks
* Refusal to participate or inability to continue participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2026-01-22 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue assessment | There will be three time points at which the measurement is assessed for both the study and the control group as follows: Pretest: At the first day Post-test 1:two weeks later . Post-test 2: four weeks later.
  Fatigue will be measured using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) scale. Higher scores indicate less fatigue.
Sleep quality | There will be three time points at which the measurement is assessed for both the study and the control group as follows: Pretest: At the first day Post-test 1: two weeks later . Post-test 2: four weeks later.
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality. A global PSQI score greater than 5 indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Haider A mohammed, PhD, Principal Investigator — Al Qadisiyah University-Faculty of Nursing
Locations (1):
- University of Baghdad, Baghdad, Iraq